CLINICAL TRIAL: NCT07217340
Title: Feasibility of a Mental-Health Intervention Based on Contemplative Sleep Practices
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Virginia (Other); Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Ken Paller, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00222189
Record Dates: First submitted 2025-09-24; First posted 2025-10-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Anxiety
Keywords: lucid dreaming; dream yoga; contemplative sleep practices; mind-body intervention; meditation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the condition of their group. They don't know if they are in the intervention study or control. The outcome assessor is blinded too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dream Yoga Inspired Intervention (Experimental): This customized contemplative training will guide participants in exploring techniques used in Tibetan Dream Yoga. Strategies in Tibetan Dream-Yoga manuals are thus transferred to a modern context and adapted as a group intervention. Goals will be set for dreaming that include gaining a degree of volitional influence over the dream. Wearable devices will be used to present cues during sleep both to provoke lucidity and to remind individuals of Dream-Yoga exercises to be engaged during sleep.
  Virtual-reality (VR) sessions provide a novel adjunct to Dream Yoga, in keeping with prior research integrating lucid dreaming and VR (Gott et al., 2021). The protocol progresses though several group activities; individuals feel themselves dispersing into a void within the VR world, and then blending with others, leading the reduced self-grasping. If this unique VR component can blur conventional self-other boundaries, it may reinforce the progressive instructions in Dream Yoga.
  Interventions: Behavioral: Dream Yoga Inspired Intervention
- Sleep Health Enhancement program (Active Comparator): A modified version of the Health Enhancement Program (HEP), which was developed as an active control condition for mindfulness-based interventions, with a particular focus on sleep hygiene. It controls for several non-specific factors such as expectations of positive change, group support, behavioural activation, facilitator attention, at-home practice, treatment duration, and format (MacCoon et al., 2012; Rosenkranz et al., 2013). Our modified HEP will be structurally equivalent to the Dream-Yoga condition, with high similarity on non-program-specific factors, including timing and number of sessions. The two VR sessions will focus on health enhancement. Participants will be taught positive health-enhancing practices, such as healthy diet and gentle exercise, with activity-based sessions covering exercise, sleep, dreaming, stress, anxiety, nutrition, journaling, music enjoyment, and drawing. Home practice and implementation of health-enhancing habits will be encouraged.
  Interventions: Behavioral: Sleep Health Enhancement program

INTERVENTIONS:
Behavioral: Dream Yoga Inspired Intervention — This customized contemplative training will guide participants in exploring techniques used in Tibetan Dream Yoga, including somatic awareness and intention-setting prior to sleep. Strategies in Tibetan Dream-Yoga manuals are thus transferred to a modern context and adapted as a group intervention. Goals will be set for dreaming that include gaining a degree of volitional influence over the dream. Participants will be instructed on how to work with their dream-world self-concept, which can include changing the environment deliberately, making other individuals appear, and switching identities with other individuals in the dream. Wearable devices will be used to present cues during sleep both to provoke lucidity and to remind individuals of Dream-Yoga exercises to be engaged during sleep. The intervention includes both wake- and sleep-based instructions, with instructions on learning to apply the new orientation in their daily lives. Participants will be contacted individually to assure
  Other Names: Contemplative Sleep Practice Intervention
  Arms: Dream Yoga Inspired Intervention
Behavioral: Sleep Health Enhancement program — The control group will receive a modified version of the Health Enhancement Program (HEP), which was developed as an active control condition for mindfulness-based interventions, with a particular focus on sleep hygiene. It controls for several non-specific factors such as expectations of positive change, group support, behavioural activation, facilitator attention, at-home practice, treatment duration, and format (MacCoon et al., 2012; Rosenkranz et al., 2013). Our modified HEP will be structurally equivalent to the Dream-Yoga condition, with high similarity on non-program-specific factors, including timing and number of sessions. The two VR sessions will focus on health enhancement. Participants will be taught positive health-enhancing practices, such as healthy diet and gentle exercise, with activity-based sessions covering exercise, sleep, dreaming, stress, anxiety, nutrition, journaling, music enjoyment, and drawing. Home practice and implementation of health-enhancing habits will
  Other Names: Health Enhancement Program
  Arms: Sleep Health Enhancement program

SUMMARY:
This is a feasibility study to test whether it is possible to deliver a program inspired by Tibetan Dream Yoga in a modern, accessible way. Dream Yoga is a set of contemplative practices that combine mental exercises during the day with techniques for becoming aware of dreaming within a dream (lucid dreaming) and engage in certain dream activities. The purpose of these practices is to help people explore and loosen rigid patterns of thought and behavior.

In this study, the investigators are developing and testing a program that includes guided imagination, meditation, and lucid-dreaming practices, supported by virtual-reality experiences and home-based sleep-monitoring technology. Participants are randomly assigned to either the Dream-Yoga-inspired program or a comparison program focused on general health and sleep education.

Because this is a feasibility trial, our main goals are to see whether people are willing and able to take part, whether they find the program acceptable, and whether the investigators can deliver it as planned. The investigators will also explore early signals of change in sleep, dreaming, and thinking.

The long-term goal of this research is to determine if such interventions could be beneficial for supporting psychological well-being, improving sleep, and enhancing creativity and flexibility of thought.

DETAILED DESCRIPTION:
Recent methodological advances enable novel scientific explorations of dreaming activities. Whereas the science of dreaming suffered historically from inadequate strategies, a new era has dawned driven by innovations in physiological sleep monitoring, two-way communication during the dream state, and lucid-dream induction.

New opportunities for dream research emerged with the demonstration that dreamers can accurately perceive spoken questions and deliver coded answers to those questions while remaining in REM sleep verified with standard polysomnography. Subsequent studies confirmed the viability of these methods and used them to explore outstanding questions about dreams. The method the experimenters use to produce lucid dreaming in the sleep laboratory, Targeted Lucidity Reactivation (TLR), was substantiated with the published demonstration that 50% of participants tested achieved a lucid dream, and now extended to the home environment based on at-home strategies previously used for slow-wave-sleep Targeted Memory Reactivation. Building on this foundation, we can use lucid-dream induction and interactive dreaming in both lab and home environments to investigate contemplative sleep practices.

Over centuries, Tibetan-Buddhist contemplatives developed and documented techniques for spiritual insight. One portrayal of insight in this context is to deconstructed conventional reality, noted that ordinary waking experience is like a dream in that people tend to grasp onto perceptual objects, thoughts, or ideas without understanding their interdependent, impermanent, and mentally constructed nature. The Buddhist literature on Dream Yoga includes manuals describing recommended practices, descriptions of benefits that can be achieved, such as enhanced cognition and emotional flexibility. The progressive exercises of Dream Yoga, including waking imagination and activities during lucid dreams, enable the dreamer to gain control over dream content, creating a platform to alter deeply ingrained habits and work to deconstruct ordinary conceptualizations.

Based on traditional wake- and sleep-based practices, we have developed an accessible strategy for personal insight, capitalizing on modern virtual-reality and sleep technology to supplement dreaming experiences. People spend a third of their lives asleep, usually oblivious to the opportunities that sleep offers. Excessive pressure in people's lives makes some consider sleep a waste of time. Yet, sleep has untapped value for mental and physical health, as increasingly acknowledged due to steady advances in the science of sleep. Today's orthodox view nevertheless holds that, although people can constructively control the context of sleep with proper habits of Sleep Hygiene, there is little control after placing a head on the pillow-sleep either goes well or it doesn't. We propose that advanced contemplative practices during sleep may hold powerful opportunities.

There is a glaring worldwide need to optimize sleep. Poor sleep is associated with many psychiatric and neurological disorders. The high prevalence of insomnia and suboptimal sleeping also contributes to other problems (e.g., low work-productivity, depression, and suicidal tendencies). A new orientation known as sleep engineering makes use of methods such as strategic sensory stimulation and sleep-and wake-based mental exercises, which can be guided by contemplative insights to enhance psychological health and well-being.

Sleep is crucial for memory, emotional regulation, and numerous aspects of health. Methods for producing transformative dream experiences and reliably provoking lucid dreaming may hold promise for reducing depression and anxiety. A randomized controlled trial was designed to test whether the intervention produces changes in sleep and waking neurophysiology, cognitive flexibility, creative insight, and self-referential focus. The intervention includes practices during dreaming and waking, whereby people learn to cultivate specific skills, aided by virtual-reality experiences and wireless sleep-technology in their own homes. As an initial step, this randomized controlled trial is designed to examine feasibility, acceptability, tolerability, and potential outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, English-speaking adults (at least 18 years old) with
* High dream recall (at least 1/month).

Exclusion Criteria:

1. a history of an established meditative practice
2. psychological or psychiatric disorders (other than mild anxiety)
3. sleep disorders, nightshift work in the past month, extreme chronotype or irregular sleeping pattern
4. use of recreational drugs in the past month
5. history of asthma, seizures or heart problems
6. unwillingness to wear headband during sleep.
7. Not having an address in the domestic United States, so residents of other countries would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Study Retention | 7 weeks (baseline to post-intervention)
  Study retention as an outcome measure will be considered positive if ≥65% of participants complete data collection at both pre- and post-intervention.
Acceptability of the Intervention | 7 weeks (throughout the intervention period)
  Acceptability will be assessed through composite measures of adherence to different elements of the intervention. The intervention will be considered acceptable if at least 70% of participants attend a minimum of five sessions. Adherence to supportive practices (dream journaling and online SHEP engagement) will also be assessed. These components will be considered acceptable if ≥75% of participants engage in Virtual Reality at a rate of ≥65%.
Tolerability of Dream Yoga Virtual Reality | 7 weeks (after each VR session)
  Tolerability will be assessed using the Simulator Sickness Questionnaire (SSQ), which measures nausea, oculomotor strain, and disorientation. The intervention will be considered tolerable if fewer than 20% of participants report severe simulator sickness or withdraw due to VR-related adverse effects. Additional safety will be monitored through adverse event logs.
Study Retention | 7 weeks (baseline to post-intervention)
  Feasibility will be assessed through study retention, defined as ≥65% of participants completing data collection at both pre- and post-intervention.

SECONDARY OUTCOMES:
Frequency of Lucid Dreaming | 7 weeks
  Lucidity will be assessed with a composite of questionnaires at week 1 and measuring changes at week 7 and using self-reports of lucid dreams recorded in daily dream journals and/or nightly reports during the 7-week intervention. The outcome will be positive if one third of participants experience at least one lucid dream.
  Self-report Questionnaires:
  1. Lucid Dreaming Skills Questionnaire (LUSK)
  2. Lucid Dream Control-Specific Experiences (LDC-SE)
Acceptability of the intervention | 7 weeks
  Acceptability will also be measured with the Acceptability of Intervention Measure (AIM), a 4-item validated scale (1-5 Likert). The intervention will be considered acceptable if the mean AIM score is ≥4.
Feasibility of the Intervention | 7 Week
  Feasibility will be measured with the Feasibility of Intervention Measure (FIM), a 4-item validated scale (1-5 Likert). The intervention will be considered feasible if the mean FIM score is ≥4 ("agree" or "completely agree").

OTHER OUTCOMES:
Change in Cognitive Flexibility Scale Score | 7 weeks (baseline to post-intervention)
  Self-report measure assessing perceived ability to shift between thoughts and adapt to changing situations.
Change in Generalized Anxiety Disorder Scale (GAD-7) Score | 7 weeks (baseline to post-intervention)
  The Generalized Anxiety Disorder Scale - 7 item (GAD-7) is a self-report questionnaire used to assess anxiety symptoms over the past two weeks. Each item is rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day"). Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Self-referential Processing: Composite od Subjective and Neural Markers | 7 weeks
  Self-referential processing will be assessed using a composite of subjective and neurophysiological measures. Subjective measures include the Mindful Attention Awareness Scale (MAAS), the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), and the Nondual Awareness Dimensional Assessment (NADA) and Beck Cognitive Insight Scale.
  Neural activity associated with self-referential processing will be indexed by frontal midline theta power (4-7 Hz) during resting-state EEG. Increased frontal midline theta has been associated with internal attention, cognitive control, and self-related processing.
  A composite score may be computed via z-score standardization or used in exploratory correlation analyses. Higher mindfulness and nondual awareness scores, together with increased frontal midline theta, will be interpreted as indicators of enhanced self-referential regulation.
Change in Probabilistic Reversal Learning Task Performance | 7 weeks
  Behavioral measure of adaptive learning and response shifting following feedback. Accuracy rate (proportion correct) and/or number of reversal errors will be assessed.
Change in Stroop Task Performance | 7 weeks
  Behavioral measure of cognitive control and interference resolution. Reaction time in milliseconds and/or accuracy will be assessed.
Change in PROMIS Anxiety Questionnaire Score | 7 weeks (baseline to post-intervention)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Questionnaire is a self-report measure assessing anxiety symptoms. It generates a T-score standardized to the general U.S. population (mean = 50, SD = 10). Higher scores indicate more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cresap Laboratory, Evanston, Illinois
  - Contemplative Sciences Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary feasibility outcomes will be shared, including retention and adherence data, responses to feasibility and acceptability questionnaires (FIM, AIM, SSQ), and basic demographic variables (age, sex). No identifying information will be included. Exploratory questionnaire data and behavioral task data may also be shared in de-identified form, depending on journal or funder requirements.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available beginning 6 months after publication of the primary results and will remain available for 5 years.

REFERENCES:
- [Background] Whitmore NW, Harris JC, Kovach T, Paller KA. Improving memory via automated targeted memory reactivation during sleep. J Sleep Res. 2022 Dec;31(6):e13731. doi: 10.1111/jsr.13731. Epub 2022 Sep 21. PMID 36129154
- [Background] Rosenkranz MA, Davidson RJ, Maccoon DG, Sheridan JF, Kalin NH, Lutz A. A comparison of mindfulness-based stress reduction and an active control in modulation of neurogenic inflammation. Brain Behav Immun. 2013 Jan;27(1):174-84. doi: 10.1016/j.bbi.2012.10.013. Epub 2012 Oct 22. PMID 23092711
- [Background] MacCoon DG, Imel ZE, Rosenkranz MA, Sheftel JG, Weng HY, Sullivan JC, Bonus KA, Stoney CM, Salomons TV, Davidson RJ, Lutz A. The validation of an active control intervention for Mindfulness Based Stress Reduction (MBSR). Behav Res Ther. 2012 Jan;50(1):3-12. doi: 10.1016/j.brat.2011.10.011. Epub 2011 Nov 11. PMID 22137364
- [Background] Konkoly KR, Appel K, Chabani E, Mangiaruga A, Gott J, Mallett R, Caughran B, Witkowski S, Whitmore NW, Mazurek CY, Berent JB, Weber FD, Turker B, Leu-Semenescu S, Maranci JB, Pipa G, Arnulf I, Oudiette D, Dresler M, Paller KA. Real-time dialogue between experimenters and dreamers during REM sleep. Curr Biol. 2021 Apr 12;31(7):1417-1427.e6. doi: 10.1016/j.cub.2021.01.026. Epub 2021 Feb 18. PMID 33607035
- [Background] Katyal S, Hajcak G, Flora T, Bartlett A, Goldin P. Event-related potential and behavioural differences in affective self-referential processing in long-term meditators versus controls. Cogn Affect Behav Neurosci. 2020 Apr;20(2):326-339. doi: 10.3758/s13415-020-00771-y. PMID 31981093
- [Background] Honma M, Plass J, Brang D, Florczak SM, Grabowecky M, Paller KA. Sleeping on the rubber-hand illusion: Memory reactivation during sleep facilitates multisensory recalibration. Neurosci Conscious. 2016;2016(1):niw020. doi: 10.1093/nc/niw020. Epub 2016 Oct 17. PMID 28184322
- [Background] Glowacki DR, Williams RR, Wonnacott MD, Maynard OM, Freire R, Pike JE, Chatziapostolou M. Group VR experiences can produce ego attenuation and connectedness comparable to psychedelics. Sci Rep. 2022 May 30;12(1):8995. doi: 10.1038/s41598-022-12637-z. PMID 35637199
- [Background] Carr, M., Konkoly, K., Mallett, R., Edwards, C., Appel, K., & Blagrove, M. (2023). Combining presleep cognitive training and REM-sleep stimulation in a laboratory morning nap for lucid dream induction. Psychology of Consciousness: Theory, Research, and Practice, 10(4), 413-430. https://doi.org/10.1037/cns0000227